CLINICAL TRIAL: NCT06412003
Title: Home-based Balance Training With Family Member Support in Adults With Multiple Sclerosis: A Feasibility Single-group Pretest-posttest Design
Brief Title: Home-based Balance Training in Adults With Multiple Sclerosis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vermont (Other)
Responsible Party: Principal Investigator, Myeongjin Bae, Principal Investigator, University of Vermont
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00002956
Record Dates: First submitted 2024-05-06; First posted 2024-05-14 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Multiple Sclerosis; Multiple Sclerosis, MS
Keywords: balance training; Home-based exercise
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Home-based balance training group (Experimental): Participants will perform the home-based balance training program for 30-40 minutes per session, 3 days per week for 12 weeks not including the two weeks of education and familiarization.
  Interventions: Behavioral: Home-based balance training

INTERVENTIONS:
Behavioral: Home-based balance training — This is a family member supported home-based balance training program designed for community-dwelling people with MS to improve balance and walking abilities as well as cognitive functions. The intervention program aims to have participants with MS reach high-intensity balance tasks during the program. A bi-weekly two-on-one, semi-structured, video-chat session with participants and their exercise supporter and research team will be conducted using videoconferencing techniques (e.g., Zoom, Skype, or Facetime).

SUMMARY:
This single-group pretest-posttest study aims to examine the feasibility domains in response to 12 weeks of home-based balance training in persons with multiple sclerosis (MS). The feasibility domains include 1) process (e.g., recruitment, attendance, adherence rate), 2) resources (e.g., total monetary costs), 3) management (e.g., assessment time), and 4) scientific outcomes (adverse events, intervention acceptability, satisfaction, treatment effects). Moreover, this study aims to evaluate physical function (i.e., balance, mobility, dual-task ability), cognitive function (i.e., cognitive processing speed, verbal memory, visuospatial memory), real-world ambulation (i.e., gait speed, gait variability, gait quantity), and self-report questionnaires (fatigue, fear of falling, walking disability, dual-tasking difficulty). Our proposed intervention is expected to deliver a feasible and accessible exercise modality for balance and cognitive improvement in persons with multiple sclerosis.

DETAILED DESCRIPTION:
Acknowledging the complex system of balance, this home-based balance training aims to address comprehensive balance control components, such as static balance, limit of stability, postural response (reactive balance), anticipatory postural transition, weight shifting, stability in gait, and stepping exercise. These balance components will be encompassed in every session to train balance function comprehensively. Exercise program will be progressed by varying sensory integrations, base of support, and simultaneous motor-cognitive tasks (i.e., dual-task).

ELIGIBILITY:
Inclusion Criteria:

* Physician-diagnosed MS
* Ages 18-75 years
* Patient Determined Disease Steps (PDDS) scale score between 2-5 (i.e., gait disability-late cane)
* Able to participate in exercise (i.e., one or fewer affirmatives on the Physical Activity Readiness Questionnaire (PAR-Q+))
* Have a webcam on a device at least the size of a full tablet (i.e., larger than a smartphone)
* Have an exercise supporter (e.g., spouse or family member) who is willing to participate in the intervention
* Not currently participating in any balance-related exercise program

Exclusion Criteria:

* Cognitively unable to read and sign informed consent form and follow verbally delivered screening assessment
* Unable to communicate in English

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility outcome: Process | From enrollment to completion of posttest (12weeks)
  This study will assess 1) recruitment rate (the number of participants screened divided by the total number of participants contacted), 2) eligibility rate (the number of participants eligible divided by total number of participants screened), 3) adherence rate (the percentages of withdrawals and completions), and 4) attendance rate (the percentages of targeted exercise sessions completed by intervention group participants who completed the study). These 4 rates will be employed to assess the feasibility of process.
Feasibility outcome: Resources | From enrollment to completion of posttest (12weeks)
  The total expenses of the study will be calculated, including materials (e.g., exercise equipment) and participant remuneration.
Feasibility outcome: Management | From enrollment to completion of posttest (12weeks)
  This study will document all videoconferencing time and baseline and follow-up assessment time. The measures will assess the time management of the intervention.
Feasibility outcome: Participant burden/satisfaction | After completion of posttest (12weeks)
  This study will assess participant burden and satisfaction through a questionnaire after the completion of the intervention. The questionnaire consists of 12 closed-ended and 2 open-ended items
Feasibility outcome: Adverse event | From enrollment to completion of posttest (12weeks)
  This study will record adverse event occurred during the intervention program.
Feasibility outcome: Intervention acceptability | From enrollment to completion of posttest (12weeks)
  This study will assess whether participants meet the prescribed exercise doses throughout the intervention program.
Feasibility outcome: exercise intensity acceptability/compliance | From enrollment to completion of posttest (12weeks)
  This study will assess whether participants adhere to a prescribed exercise intensity dose throughout the intervention program. An exercise log will be employed to assess exercise intensity acceptability.

SECONDARY OUTCOMES:
Changes in balance as measured by Timed Up and Go/Dual-task Timed Up and Go | Baseline and after completion of an intervention (12weeks)
  The Timed Up and Go test assesses mobility, anticipatory postural control, and dynamic balance. Dual-task Timed Up and Go will assess cognitive-motor interference
Changes in functional mobility as measured by 5-time sit-to-stand | Baseline and after completion of an intervention (12weeks)
  The test is a valid measure of functional mobility and dynamic balance performance in people with multiple sclerosis.
Changes in static balance as measured by4-stage static balance tests | Baseline and after completion of an intervention (12weeks)
  The test assesses static balance ability in participants with multiple sclerosis.
Changes in cognitive function as measured by Brief International Cognitive Assessments for MS (BICAMS) | Baseline and after completion of an intervention (12weeks)
  This neuropsychological cognitive test battery is a valid measure for persons with multiple sclerosis. The BICAMS includes Symbol Digit Modalities Test (SDMT), California Verbal Learning Test (CVLT2), and revised Brief Visuospatial Memory Test (BVMTR), whose tests primarily target to measure cognitive processing speed, verbal memory, and visuospatial memory, respectively.
Changes in community mobility perception as measured by Environmental Analysis of Mobility Questionnaire (EAMQ) | Baseline and after completion of an intervention (12weeks)
  This study will assess perceptions of community mobility in relation to specific environmental situations or tasks using the Environmental Analysis of Mobility Questionnaire (EAMQ). EAMQ consists of 24 items grouped within 8 environmental dimensions: distance, temporal, ambient, terrain, physical load, postural transition, attention, and density. Participants will be asked to rate the frequency of avoidance of specific mobility tasks on a 5-point scale ranging from 1 (never avoid) to 5 (always avoid). Total scores for each dimension will be calculated and assessed in the analyses.
Changes in fear of falling as measured by Fall Efficacy Scale-International (FES-I) | Baseline and after completion of an intervention (12weeks)
  This survey assesses how concerned one is about falling during both physical and social activities. Participants will be asked to rate 16 items using a 4-point Likert-type scale (1=not at all concerned, 4=very concerned), with lower scores indicating less concern about falling.
Changes in self-reported walking disability as measured by Multiple Sclerosis Walking Scale-12v2 (MSWS-12v2) | Baseline and after completion of an intervention (12weeks)
  The Multiple Sclerosis Walking Scale-12v2 (MSWS-12v2) will assess perceived limitations to their walking under varying conditions. The survey includes 12 items, of which three items are rated on a 3-point scale (1= not at all, 2=sometime, 3=a lot) and nine items by a 5-point scale (1=not limited, 5=extremely limited). Total scores range from 12 to 54, with higher scores indicating greater perceived mobility impairment.
Changes in self-reported dual-tasking difficulty as measured by Dual-task Impact on Daily-Living Activities Questionnaire (DIDA-Q) | Baseline and after completion of an intervention (12weeks)
  The Dual-task Impact on Daily-Living Activities Questionnaire (DIDA-Q) contains 16 items rated on 5-point Likert-type scale (0=no difficulty, 4=extremely difficult). A total score ranges from 0 to 76, with higher scores demonstrating greater difficulty in dual-tasking.
Changes in self-reported fatigue as measured by Fatigue Scale for Motor and Cognitive Functions (FSMC) | Baseline and after completion of an intervention (12weeks)
  This survey consists of 20 items, including 10 items for motor fatigue and 10 items for cognitive fatigue, with scales ranging from 1 (i.e., does not apply at all) to 5 (i.e., applies completely). Higher score indicates greater level of fatigue.
Changes in Real-world ambulation metrics as measured by tri-axial accelerometer | Baseline and after completion of an intervention (12weeks)
  The AX3 3-axis accelerometer (Axivity, York, UK) will be employed to collect real-world ambulation, including gait speed and stride regularity.
Changes in exercise intention | Baseline and after completion of an intervention (12weeks)
  The questionnaire will assess exercise supporters' attitudes, perceived behavioral control, and intentions by a constructed questionnaire based on the theory of planned behavior. The questionnaire includes 61 items, with a higher score indicating greater exercise support attitudes, perceived behavioral control, and intentions

REFERENCES:
- [Derived] Bae M, Gell NM, Ramsey C, Kasser SL. Feasibility of home-based high-intensity balance training in persons with multiple sclerosis: A pretest-posttest study. Clin Rehabil. 2026 Jan;40(1):30-43. doi: 10.1177/02692155251384079. Epub 2025 Oct 17. PMID 41105745